CLINICAL TRIAL: NCT03371056
Title: Innovative Strategies for Perinatal Infectious Risk Reduction
Brief Title: Maternal- Fetal Infection
Acronym: InSPIRe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bforcure (Unknown); BPIfrance (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: K170907J
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Neonatal Infection
Keywords: Neonatal infections; maternal-fetal infection; group B streptococcus; vaginal sample; antibiotic prophylaxis; bacterial resistance

STUDY DESIGN:
Intervention Model Description: There are 4 pre-specified groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Woman at low risk of infection (Experimental): Women with systematic vaginal sample for detection of GBS will be included.
  Interventions: Biological: Bacteriological analyses on clinical samples performed with swabs
- Woman with high risk of infection > 37 SA (Experimental): Women with premature rupture of membranes (> 12 hours before labor) but > 37 SA will be included.
  Interventions: Biological: Bacteriological analyses on clinical samples performed with swabs
- Women with premature rupture of membranes (<37SA) (Experimental): Woman with high risk of infection <37SA
  Interventions: Biological: Bacteriological analyses on clinical samples performed with swabs
- Women with premature delivery or premature delivery threat (Experimental): Woman with high risk of infection <37SA and Women with premature delivery or premature delivery threat
  Interventions: Biological: Bacteriological analyses on clinical samples performed with swabs

INTERVENTIONS:
Biological: Bacteriological analyses on clinical samples performed with swabs — Bacteriological analyses will be performed to assess the InSPIRe kit

SUMMARY:
The purpose of the protocol is to validate a novel point of care multiplex system to detect and characterize microorganisms responsible for neonatal sepsis, as well as biomarkers of infection, from a simple vaginal sample, in order to improve the prevention of perinatal bacterial infections.

DETAILED DESCRIPTION:
Early-onset neonatal sepsis (EOS) is a major global public health challenge. Prevention during pregnancy and delivery, early diagnosis and treatment of perinatal infections are essential to avoid EOS. Risk factors for include prematurity, maternal Group B streptococcus (GBS) colonization, premature rupture of membranes (PROM), and chorioamnionitis. Screening and intrapartum antimicrobial prophylaxis administered to GBS-colonized women has reduced early onset GBS infections. However, other pathogens are frequently involved in EOS following preterm PROM and preterm birth (PTB), such as Gram-negative bacteria and Staphylococci, which are not covered by penicillin prophylaxis. The prevalence of neonatal infection arising from antibiotic-resistant bacteria is increasing, thus the challenge is to eliminate the widespread unnecessary use of broad-spectrum antibiotics to treat non-infected infants, while recognizing when antibiotics are truly needed. Rapid diagnostic test(s) to detect and quantify specifically pathogens in vaginal samples, could be a major breakthrough. Several rT- PCR ( reverse Transcriptase Polymerase Chain Reaction) tests are on the market, however so far no test is able to detect, quantify and characterize in terms of antibiotic resistance and virulence genes, a range of pathogens.

A novel multiplex platform, using microfluidics technology, is under development by Elvesys, Inc in France. This platform will be able to offer results within 15 minutes on-site.

In addition, the study of the vaginal microbiome may identify signatures associated with a risk of maternal-fetal infection, particularly in case of PROM or PTB. Advanced sequencing technology and metagenomics will be used to characterize these signatures, and may lead to further markers to be included in the point-of-care test. Finally, biomarkers of inflammation will be detected, including IL-6 (Interleukin).

In this study, the InSPIRe platform will be compared in the laboratory to conventional microbiological and immunological detection.

Four groups of pregnant women will be recruited in prospective cohorts : uneventful pregnancies, term PROM, preterm labor and preterm PROM.

The purpose of the InSPIRe project is to improve the prevention of perinatal bacterial infections, with the novel Elvesys point of care system to rapidly detect and characterize microorganisms responsible for neonatal sepsis from a single vaginal sample.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman,
* Gestational age over 22 SA,
* Patient agreeing to sign informed consent,
* Patient aged at least 18 years old,
* Patient with health insurance,
* Singleton, twin or multiple pregnancy.

Exclusion Criteria:

* Fetal death or non-viable fetus,
* maternal age under 18,
* Patient unable to express her consent,
* Patient under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Presence of Streptococcus B | Day 0
Presence of Streptococcus B | until 20 weeks

SECONDARY OUTCOMES:
Maternal fetal infection | until 20 weeks + 3 days
  Infection is proved if at least a sample, generally sterile, is positive to a germ in association with a positive clinical, biological or radiologic sign of infection such as C-reactive protein or chest radiography.
A positive bacteriological result in the vaginal sample | Day 0
  A positive result is defined as the presence of one of the subsequent germ in the bacteriological culture:
  * Escherichia coli (E. coli)
  * Streptococcus pneumoniae,
  * Group A Streptococcus
  * Haemophilus ssp (influenzae, parainfluenzae)
  * Staphylococcus aureus
  * Streptococcus milleri group
  * Enterococcus faecalis
  * Other Gram-negative bacilli type enterobacteria (Klebsiella pneumonia, Proteus mirabilis)
  * Anaerobics (Prevotella sp, bacteroid fragilis)
A positive bacteriological result in the vaginal sample | until 20 weeks
  A positive result is defined as the presence of one of the subsequent germ in the bacteriological culture:
  * Escherichia coli (E. coli)
  * Streptococcus pneumoniae,
  * Group A Streptococcus
  * Haemophilus ssp (influenzae, parainfluenzae)
  * Staphylococcus aureus
  * Streptococcus milleri group
  * Enterococcus faecalis
  * Other Gram-negative bacilli type enterobacteria (Klebsiella pneumonia, Proteus mirabilis)
  * Anaerobics (Prevotella sp, bacteroid fragilis)
Vaginal dysmorphism | day 0
  Defined by lactobacillus's decrease or loss in association with the spread of anaerobic flora.
Vaginal dysmorphism | until 20 weeks
  Defined by lactobacillus's decrease or loss in association with the spread of anaerobic flora.
Antibiotic resistance | Day 0
  Highlighted by a resistant profile in bacteriological culture for various classes of antibiotics such as β-lactamines, macrolides or aminoamides.
Antibiotic resistance | until 20 weeks
  Highlighted by a resistant profile in bacteriological culture for various classes of antibiotics such as β-lactamines, macrolides or aminoamides.
Highlighting specific virulence markers | Day 0
  Like GBS clone CC17, Enterobacteriaceae that produce capsular antigen type K1. By usual molecular techniques.
Highlighting specific virulence markers | until 20 weeks
  Like GBS clone CC17, Enterobacteriaceae that produce capsular antigen type K1. By usual molecular techniques.
Maternal local biomarkers definition | Day 0
  Presence or lack of RNA sequences and/or human specific protein detected by RT-PCR or ELISA-PCR depending on the presence or lack of a proved or suspected maternal fetal infection.
Maternal local biomarkers definition | until 20 weeks
  Presence or lack of RNA sequences and/or human specific protein detected by RT-PCR or ELISA-PCR depending on the presence or lack of a proved or suspected maternal fetal infection.
Bacteriological signature definition | Day 0
  Presence or lack of specific bacteriological sequences detected by global sequencing and metagenomics analyses
Bacteriological signature definition | until 20 weeks
  Presence or lack of specific bacteriological sequences detected by global sequencing and metagenomics analyses
Chorioamnionitis | Day 0
  Clinical or paraclinical factors associated with risk of chorioamnionitis or maternal fetal infection such as prematurity, clinical signs (maternal fever, fetal tachycardia, increase in C-reactive protein, hyperleukocytosis, pus-like amniotic fluid) , oligohydramnios (defined by the greatest cistern < 25 mm); increase in pro-calcitonin in umbilical cord ok histological signs of placental inflammation.
  Clinical chorioamnionitis is defined as a maternal fever> 39° (in one shot) with no other cause or >38°(confirmed) in association with abnormal fetal heartbeat (>160/min exceeding 10 min), maternal hyperleukocytosis (>15000/mm3 without corticotherapy) or pus-like amniotic fluid.
  Histological chorioamnionitis is defined by the presence of neutrophil polynuclears in amnion or chorion in association with the presence of neutrophil polynuclears in umbilical cord blood vessels.
Chorioamnionitis | until 20 weeks
  Clinical or paraclinical factors associated with risk of chorioamnionitis or maternal fetal infection such as prematurity, clinical signs (maternal fever, fetal tachycardia, increase in C-reactive protein, hyperleukocytosis, pus-like amniotic fluid) , oligohydramnios (defined by the greatest cistern < 25 mm); increase in pro-calcitonin in umbilical cord ok histological signs of placental inflammation.
  Clinical chorioamnionitis is defined as a maternal fever> 39° (in one shot) with no other cause or >38°(confirmed) in association with abnormal fetal heartbeat (>160/min exceeding 10 min), maternal hyperleukocytosis (>15000/mm3 without corticotherapy) or pus-like amniotic fluid.
  Histological chorioamnionitis is defined by the presence of neutrophil polynuclears in amnion or chorion in association with the presence of neutrophil polynuclears in umbilical cord blood vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mandelbrot, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Claire Poyart, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Pierre Yves Ancel, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hopital Louis Mourier, Colombes
  - Hôpital Cochin, Paris
  - Hopital Bichat, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joubrel C, Tazi A, Six A, Dmytruk N, Touak G, Bidet P, Raymond J, Trieu Cuot P, Fouet A, Kerneis S, Poyart C. Group B streptococcus neonatal invasive infections, France 2007-2012. Clin Microbiol Infect. 2015 Oct;21(10):910-6. doi: 10.1016/j.cmi.2015.05.039. Epub 2015 Jun 5. PMID 26055414
- [Background] Dussaux C, Senat MV, Bouchghoul H, Benachi A, Mandelbrot L, Kayem G. Preterm premature rupture of membranes: is home care acceptable? J Matern Fetal Neonatal Med. 2018 Sep;31(17):2284-2292. doi: 10.1080/14767058.2017.1341482. Epub 2017 Jul 6. PMID 28612662
- [Background] Kayem G, Batteux F, Girard N, Schmitz T, Willaime M, Maillard F, Jarreau PH, Goffinet F. Predictive value of vaginal IL-6 and TNFalpha bedside tests repeated until delivery for the prediction of maternal-fetal infection in cases of premature rupture of membranes. Eur J Obstet Gynecol Reprod Biol. 2017 Apr;211:8-14. doi: 10.1016/j.ejogrb.2017.01.013. Epub 2017 Jan 12. PMID 28160689
- [Background] Lorthe E, Ancel PY, Torchin H, Kaminski M, Langer B, Subtil D, Sentilhes L, Arnaud C, Carbonne B, Debillon T, Delorme P, D'Ercole C, Dreyfus M, Lebeaux C, Galimard JE, Vayssiere C, Winer N, L'Helias LF, Goffinet F, Kayem G. Impact of Latency Duration on the Prognosis of Preterm Infants after Preterm Premature Rupture of Membranes at 24 to 32 Weeks' Gestation: A National Population-Based Cohort Study. J Pediatr. 2017 Mar;182:47-52.e2. doi: 10.1016/j.jpeds.2016.11.074. Epub 2017 Jan 9. PMID 28081890
- [Background] Delorme P, Goffinet F, Ancel PY, Foix-L'Helias L, Langer B, Lebeaux C, Marchand LM, Zeitlin J, Ego A, Arnaud C, Vayssiere C, Lorthe E, Durrmeyer X, Sentilhes L, Subtil D, Debillon T, Winer N, Kaminski M, D'Ercole C, Dreyfus M, Carbonne B, Kayem G. Cause of Preterm Birth as a Prognostic Factor for Mortality. Obstet Gynecol. 2016 Jan;127(1):40-48. doi: 10.1097/AOG.0000000000001179. PMID 26646125
- [Background] Plainvert C, El Alaoui F, Tazi A, Joubrel C, Anselem O, Ballon M, Frigo A, Branger C, Mandelbrot L, Goffinet F, Poyart C. Intrapartum group B Streptococcus screening in the labor ward by Xpert(R) GBS real-time PCR. Eur J Clin Microbiol Infect Dis. 2018 Feb;37(2):265-270. doi: 10.1007/s10096-017-3125-2. Epub 2017 Oct 29. PMID 29082442
- [Background] Six A, Firon A, Plainvert C, Caplain C, Bouaboud A, Touak G, Dmytruk N, Longo M, Letourneur F, Fouet A, Trieu-Cuot P, Poyart C. Molecular Characterization of Nonhemolytic and Nonpigmented Group B Streptococci Responsible for Human Invasive Infections. J Clin Microbiol. 2016 Jan;54(1):75-82. doi: 10.1128/JCM.02177-15. Epub 2015 Oct 21. PMID 26491182